CLINICAL TRIAL: NCT03741907
Title: French Ambulatory and Misgav Ladach Cesarean Section Techniques : a Results of a Comparative Randomized Trial.
Brief Title: Comparing French Ambulatory and MISGAV-LADACH C-Section Techniques
Acronym: MLC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Tunis El Manar (Other)
Responsible Party: Principal Investigator, Kaouther Dimassi, Associate professor, University Tunis El Manar
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: FAUCS MongiSlim
Record Dates: First submitted 2018-11-05; First posted 2018-11-15 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Cesarean Section
Keywords: Cesarean; Surgery; Birth; Recovery; Outcomes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FAUCS (Experimental): French Ambulatory C-section
  Interventions: Procedure: FAUCS
- MLC (Active Comparator): Gold Standard
  Interventions: Procedure: MLC

INTERVENTIONS:
Procedure: FAUCS — extraperitoneal cesarean with a paramedian left section
  Other Names: French Ambulatory Cesarean section
  Arms: FAUCS
Procedure: MLC — Gold standard
  Other Names: "Misgav Ladach" Method
  Arms: MLC

SUMMARY:
In the last decades cesarean section rates are getting higher in many countries. The rise in those rates encourages obstetricians to improve operative techniques for a better maternal and fetal outcome.

Despite its worldwide spread, a general consensus on the most appropriate technique to use has not yet been reached.

The most known surgical technique is the MLC . A modified extraperitoneal method of caesarean section :" French Ambulatory Cesarean Section ( FAUCS) was described in the middle of the 90's by "Denis Fauck" and "Jacques Henri Ravina " However, no study comparing these two cesarean techniques was conducted. From where the investigators initiate this study .

DETAILED DESCRIPTION:
Caesarean Section (CS) is one of the most commonly performed operations worldwide The rate of CS continues to rise, despite initiatives to counter this trend. Cesarean sections have a higher morbidity rate than vaginal deliveries, with a substantial care and cost measurable by the mean hospital stay, the use of analgesics, and the potential for complications . Crucially, the birth of a new baby is an unique incentive to return quickly to "normal" function. Improving the cesarean section techniques is therefore of considerable importance in modern obstetrics.

One of the most widely used cesarean section techniques is the MLC method developed by Michael Stark et al. This approach is indicated as the optimal technique in view of its characteristic of reducing lower pelvic discomfort and pain, thus improving quality of life However, this intraperitoneal C-section interfere at least with future fertility desire.

The French Ambulatory Cesarean Section (FAUCS) technique has been employed by 10 practitioners in France for approximately 20 years. In a retrospective study over 3000 cases this innovative approach seems to provide a shorter recovery time with a Hospital discharge the day after surgery . Investigators introduced this technique in "Mongi Slim" university hospital in January 2018. In this study, investigators compare the FAUCS and the MLC techniques in termes of mother and child outcomes

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy
* gestational age of at least 37 weeks of amenorrhea
* indication of elective cesarean delivery mode (breech presentation ; Fetal macrosomia ; Placenta previa)

Exclusion Criteria:

* Fetal pathology diagnosed prenatally( intrauterine growth restriction , malformation, genetic pathology ... )
* Morbidity adherent placenta
* emergency Cesarean section

Ages: 18 Years to 48 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2018-08-27 (Actual); Primary Completion 2019-03-20 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
changes in post operative pain | 6 hours ; 12 hours , 18 hours , 24 hours
  changes in postoperative analgesic requirements, changes in self reported pain using the Visual Analog Scale for Pain (VAS Pain) intensity ( The pain VAS is a single-item scale.For pain intensity, the scale is most commonly anchored by "no pain" (score of 0) and "pain as bad as it could be" or "worst imaginable pain" (score of 100 [100-mm scale] )
delay to hospital discharge | up to 72 hours
  report of total days spent in hospital after surgery

SECONDARY OUTCOMES:
blood loss | the day before surgery and the day after surgery (24 hours)
  change in hemoglobin and hematocrit rate
operation time | during the surgery
  total operation time ; time to fetal extraction ; time to uterine sutures
rate of short term incidents | during the surgery and 24 hours after surgery
  rate of hemorrhage, rate of transfusion, rate of bladder injury
patient autonomy questionnaire | up to 48 hours after surgery
  time to first spontaneous miction, time to stand up ; time to first complete meal, time to first breastfeeding
newborn overall condition | 5 minutes from birth
  Apgar score ( The Apgar score is determined by evaluating the newborn baby on five simple criteria on a scale from zero to two, then summing up the five values thus obtained. The resulting Apgar score ranges from zero to 10. The five criteria are summarized using words chosen to form an ackronym (Appearance, Pulse, Grimace, Activity, Respiration).he test is generally done at 1 and 5 minutes after birth and may be repeated later if the score is and remains low. Scores 7 and above are generally normal; 4 to 6, fairly low; and 3 and below are generally regarded as critically low and cause for immediate resuscitative efforts.)
neonatal acid base balance | immediately after fetal extraction
  Cord blood gases

CONTACTS AND LOCATIONS:
Overall Officials: kaouther dimassi, MD, Principal Investigator — University Tunis El Manar , Faculty of medicine Tunis
Locations (1):
- Kaouther Dimassi, Tunis, Sidi Daoued La Marsa, Tunisia

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-05): https://cdn.clinicaltrials.gov/large-docs/07/NCT03741907/Prot_SAP_000.pdf